CLINICAL TRIAL: NCT03320967
Title: COpeptin in Critically Ill Paediatric and Neonatal Intensive Care Patients and Its Association With Arterial Hypotension. A Single-centre Prospective Observational Study.
Brief Title: Copeptin and Arterial Hypotension in Critically Ill Paediatric and Neonatal Intensive Care Patients
Acronym: COPNIC
Status: Completed | Type: Observational
Sponsor: Vincenzo Cannizzaro (Other)
Responsible Party: Sponsor-Investigator, Vincenzo Cannizzaro, Vice-head Department of Pediatric Intensive Care and Neonatology, University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Other Study IDs: KISPI-COPNIC
Record Dates: First submitted 2017-10-04; First posted 2017-10-25 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Arterial Hypotension in Critically Ill Neonatal and Pediatric Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Copeptin in plasma — Copeptin will be measured in EDTA-Plasma. Samples will be stored for batch analyses later.

SUMMARY:
Blood copeptin will be measured during the routine treatment of neonates, children and adolescents on the Intensive Care Unit of the University Children's Hospital Zurich at different time points (admission, 12, 24, 48, 96, 168 hours after admission). These values will be primarily analysed for their variability and their association with arterial hypotension. Blood samples will be drawn together with otherwise medically indicated blood withdrawals to avoid extra harm. Further, copeptin values will be compared to clinical and vital parameters, all of them open-label available during clinical routine. Copeptin's predictive value for patients' outcome will be analysed as secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age: first day of life until 18th birthday.
* Ability of the care taker or the adolescent (if≥14 years of age) to understand verbal and written instructions and informed consent in German.

Exclusion Criteria:

* Care taker or adolescent (if ≥14 years of age) unwilling to give written informed consent.
* Care taker or adolescent (if ≥14 years of age) not understanding German and without a family member able to translate.
* Adolescent (if ≥14 years of age) unwilling to give written informed consent following sedation < 24 hours.
* Care takers of long-term sedated (>24 hours) adolescents (if ≥14 years of age) unwilling to give written informed consent or not present within 24 hours.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a study designed to explore Copeptin values in all kinds of critically ill paediatric patients. Patients with normal blood pressures will allow calculating Copeptin reference values for the ones requiring cardiovascular support. Therefore, all patients, irrespective of their medical condition (e.g. medical or surgical, mildly or severely affected) and their age (neonates to adolescents) admitted to the Intensive Care Unit of the University's Children Hospital Zurich will be eligible, as long as they fulfil the mentioned inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Blood copeptin in arterial normo- and hypotension | Up to 168 hours.
  Average change of blood copeptin in patients with both arterial normo- and hypotension and different pathologies.

SECONDARY OUTCOMES:
Length of stay on the intensive care unit | Up to 168 hours.
  Association of copeptin values with length of stay on the intensive care unit.
Length of respiratory support | Up to 168 hours.
  Association of copeptin values with length of respiratory Support.
Length and dose of catecholamine therapy | Up to 168 hours.
  Association of copeptin values with length and dose of catecholamine therapy.
Rate of death | Up to 168 hours.
  Rate of death at 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Vinzenco Cannizzaro, MD, PhD, Study Director — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT03320967/Prot_000.pdf